CLINICAL TRIAL: NCT05428956
Title: A Randomized Controlled Trial of Two Inhalation Methods Using a Pressurized Metered Dose Inhaler With Valved Holding Chamber to Assess Improvement in Lung Function After Short-acting Beta-2 Agonist Administration in Treatment-naïve Adult Patients With Bronchial Asthma
Brief Title: Two Inhalation Methods Using a Pressurized Metered Dose Inhaler With Valved Holding Chamber to Assess Improvement in Lung Function After SABA Administration in Bronchial Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Inderpaul singh, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: INT/IEC/2016/976
Record Dates: First submitted 2022-06-15; First posted 2022-06-23 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: All the patients will receive inhaled salbutamol using two techniques during lung function testing on two successive days. Patient will be randomized 1:1 to receive inhaled salbutamol by performing either a single breath holding maneuver or by five tidal breaths on the first day of evaluation. Each patient will undergo spirometry using the other alternative procedure on the next day. The randomization sequence will be computer generated. The sequence generated will be kept in a sealed opaque envelope and will be opened at the time of procedure
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will perform the spirometry after use of short acting bronchodilator with a spacer using both single breath and 5-tidal breath on two consecutive days. The investigator, care provider and outcome assessor will be masked for allocation. The spirometry will be performed by a respiratory technician not involved in patient care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single breath technique (Active Comparator): The technique of single maximal inhalation will be demonstrated to all the patients by a technician. In brief the patient will be asked to inhale slowly and maximally and hold the breath for at least 5 seconds. After the breath holding maneuver the patient will be asked to exhale. Salbutamol (100µg) be administered in a dose of 2 puffs, each after a one minute interval. The duration of the breath hold will be measured by a stop watch.
  Interventions: Procedure: Single Inhalation technique; Procedure: Tidal inhalation technique
- Tidal breath technique (Experimental): The technique of 5 tidal breaths will be demonstrated to all the patients by a technician. In brief the patient will be asked to inhale 5 tidal breaths after administrating salbutamol in the spacer. After each breath patient will be asked to breathe out in the spacer. The spacer has a one way-valve and does not allow the exhaled air to enter in to the chamber, thus preventing rebreathing and dilution of the inhaled medicine. Salbutamol (100µg) be administered in a dose of 2 puffs, each after a one minute interval
  Interventions: Procedure: Single Inhalation technique; Procedure: Tidal inhalation technique

INTERVENTIONS:
Procedure: Single Inhalation technique — Single maximal inhalation with breath hold technique
Procedure: Tidal inhalation technique — 5 tidal breaths technique

SUMMARY:
Bronchial asthma is a chronic inflammatory disorder characterized by recurrent reversible episodes of breathlessness, wheezing, chest tightness and/ or cough. The prevalence of asthma in India is about 2%, and asthma is responsible for significant morbidity. A diagnosis of asthma is made in the presence of clinical symptoms with or without reversibility on spirometry assessment.1 Treatment comprises of inhaled medications that are used either as controller medication or a reliever medications.

In a recent study involving asthmatic children, single maximal inhalation with breath hold was not found to be superior to tidal breathing for improvement in peak expiratory flow rates.

The authors hypothesized that both the techniques would improve FEV1 similarly.

DETAILED DESCRIPTION:
Bronchial asthma is a chronic inflammatory disorder characterized by recurrent reversible episodes of breathlessness, wheezing, chest tightness and/ or cough.1 The prevalence of asthma in India is about 2%, and asthma is responsible for significant morbidity. A diagnosis of asthma is made in the presence of clinical symptoms with or without reversibility on spirometry assessment.1 Treatment comprises of inhaled medications that are used either as controller medication or a reliever medications.1 PEF measurements are known to be affected by the technique and the equipment by which it is measured, and thus proper instructions and training are essential for the patient.1 PEF measurements have been used in the past as a surrogate to FEV1 measurements, but the correlation between them is poor and hence they should not be used interchangeably. If PEF falls below 80% of personal best, it is suggestive of inadequate disease control.1 Inhaled medications are delivered through various device either as dry powder forms or in a pressurized meter dose inhaler (pMDI). However, the drug delivery is variable and a pMDI delivers only 10-20% of the nominal dose per actuation or puff, even when used correctly.2,3 Use of spacer improves the drug delivery and the recent Indian guidelines recommends use of pMDI with a spacer as an effective drug delivery system. Tidal breathing with a pMDI with spacer is as effective as the single breath method as per the British/Scottish Intercollegiate Guidelines Network (SIGN) recommendations.4 Breath-holding is usually recommended after the aerosol inhalation, but there is limited information on the clinical importance of breath-holding in adult asthmatic patients. In a recent study involving asthmatic children, single maximal inhalation with breath hold was not found to be superior to tidal breathing for improvement in peak expiratory flow rates.5 Information on comparative efficacy of either method is limited in adult asthmatics. The authors hypothesized that both the techniques would improve FEV1 similarly. Thus, the objective of the present study is to assess improvement in lung function (FEV1) after short-acting beta-2 agonist administration in treatment-naïve adult patients with bronchial asthma with a single maximal inhalation with breath-hold versus 5 tidal breaths during inhalation using a valved holding chamber.

ELIGIBILITY:
Inclusion Criteria:

(a) Patients with a physician diagnosis of bronchial asthma undergoing spirometry (b) ability to provide informed consent to participate in the study

Exclusion Criteria:

(a) Patients having active pulmonary tuberculosis; (b) pregnancy; (c) patients already on inhaled or oral bronchodilators or corticosteroids as part of asthma treatment; and, (d) failure to provide informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 897 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change in FEV1 (ml) | 48 hours
  absolute change in FEV1 after inhaled salbutamol administered with a valved spacer using single maximal inhalation with breath hold and 5-tidal breaths technique.

SECONDARY OUTCOMES:
percentage change in FEV1 | 48 hours
  percentage change in FEV1 after inhaled salbutamol administered with a valved spacer using single maximal inhalation with breath hold and 5-tidal breaths technique
Change in FVC in mL | 48 hours
  absolute change in FVC, and PEFR after inhaled salbutamol administered with a valved spacer using single maximal inhalation with breath hold and 5-tidal breaths technique
percentage change in FVC | 48 hours
  percentage change in FVC after inhaled salbutamol administered with a valved spacer using single maximal inhalation with breath hold and 5-tidal breaths technique
percentage change in PEFR | 48 hours
  percentage change in PEFR after inhaled salbutamol administered with a valved spacer using single maximal inhalation with breath hold and 5-tidal breaths technique
Change in PEFR, in mL | 48 hours
  absolute change in PEFR after inhaled salbutamol administered with a valved spacer using single maximal inhalation with breath hold and 5-tidal breaths technique

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Bronchoscopy suite, PGIMER, Chandigarh
  - Chest clinic, Chandigarh

IPD SHARING:
Plan to Share IPD: Undecided
Will share IPD on request